

#### **Statistical Analysis Plan**

 Study Code
 PT010010

 NCT #
 NCT03075267

 Version
 Ver. 1.0

 Date
 24 August 2017

A Phase I, Randomized, Double-Blind, Parallel-Group Study to Assess the Pharmacokinetics and Safety of Two Doses of PT010 and a Single Dose of PT003 in Healthy Chinese Adult Subjects Following A Single Administration and After Chronic Administration for 7 Days

Protocol Nos.: PT010010 Date: 24 Aug 2017 

## STATISTICAL ANALYSIS PLAN FOR STUDY PT010010

**Protocol Number:** PT010010

Investigational Drug and Drug Number:

BGF MDI; PT010

GFF MDI; PT003

**Indication:** COPD

**Dosage Form/Dose:** • BGF MDI 320/14.4/9.6 μg ex-actuator

• BGF MDI 160/14.4/9.6 μg ex-actuator

• GFF MDI 14.4/9.6 μg ex-actuator

**PT010010 Protocol Title:** A Phase I, Randomized, Double-Blind, Parallel-Group, Study to Assess the Pharmacokinetics and Safety of Two Doses of PT010 and a Single Dose of PT003 in Healthy Chinese Adult Subjects Following A Single Administration and After Chronic Administration for 7 Days

**Date of Issue:** 24 Aug 2017

**Version:** Version 1.0



Statistical Analysis Plan Protocol Nos.: PT010010 Date: 24 Aug 2017 

## Signed Agreement on Statistical Analysis Plan

## FINAL SIGN-OFF SIGNATURES

| Primary Biostatistician<br>and Peer Reviewer: |
|-----------------------------------------------|
| Author: |
| Co-Author: |
| Approved by: |
| Approved by: |

Pearl

Statistical Analysis Plan Protocol Nos.: PT010010 Date: 24 Aug 2017 

| Approved by: |
|--------------|
| a |
| Approved by: |
| 8 |



Statistical Analysis Plan Protocol Nos.: PT010010 Date: 24 Aug 2017 

| Change Log | | | |
|-------------|----------------|----------------------------------|------------|
| Version No. | Effective Date | Reason for the Change / Revision | Supersedes |

Protocol Nos.: PT010010 Date: 24 Aug 2017 

#### **TABLE OF CONTENTS**

| 1. | INT | RODUCTION | 12 |
|---|---|---|---|
| 2. | STU | DY OBJECTIVES AND ENDPOINTS | 12 |
| | 2.1 | STUDY OBJECTIVES | 12 |
| | 2.1 | 2.1.1 Primary Objective | |
| | | 2.1.2 Secondary Objective | |
| | 2.2 | STUDY ENDPOINTS | |
| | | 2.2.1 Pharmacokinetic Endpoint | |
| | | 2.2.2 Secondary Endpoint. | |
| 3. | STU | DY DESIGN AND ANALYTICAL CONSIDERATIONS | |
| | 3.1 | STUDY DESIGN | 13 |
| | 0.1 | 3.1.1 Overall Study Design and Plan | |
| | | 3.1.2 Prior, Concomitant, Post-Treatment, Prohibited Medications, and Other Restrictions | |
| | | 3.1.2.1 Surgical Procedure/Intervention Restrictions | |
| | | 3.1.2.2 Dietary Restrictions | |
| | | 3.1.2.3 Illicit Drugs and/or Drugs of Abuse Restriction | |
| | | 3.1.2.4 Smoking Restrictions | |
| | 3.2 | RANDOMIZATION AND BLINDING | |
| | 3.3 | HYPOTHESIS TESTING | |
| | 3.4 | INTERIM ANALYSIS | 17 |
| | 3.5 | SAMPLE SIZE | 17 |
| | 3.6 | STUDY PROCEDURES | 17 |
| | 3.7 | SCHEDULE OF ASSESSMENTS. | 17 |
| 4. | DAT | TA AND ANALYTICAL QUALITY ASSURANCE | 17 |
| 5. | ANA | ALYSIS POPULATIONS | 17 |
| | 5.1 | POPULATION DEFINITIONS | 17 |
| | 5.1 | 5.1.1 Safety Population | |
| | | 5.1.2 Pharmacokinetic (PK) Population | |
| | 5.2 | Populations for Analyses | |
| 6. | | CIFICATION OF ENDPOINTS AND VARIABLES | |
| 0. | 6.1 | DEMOGRAPHICS AND BASELINE CHARACTERISTICS | |
| | 6.2 | PHARMACOKINETICS | |
| | 6.3 | SAFETY ASSESSMENTS | |
| | 0.3 | 6.3.1 Physical Examination | |
| | | 6.3.2 Vital Signs | |
| | | 6.3.3 12-Lead Electrocardiogram | |
| | | 6.3.4 Clinical Laboratory Tests | |
| | | 6.3.5 Adverse Events | |
| | | 6.3.6 Urine Drug Screening/Alcohol Breath Testing. | |
| | | 6.3.7 Pregnancy Test | |
| | | 6.3.8 Concomitant Medications/Treatments | |
| 7. | STA | TISTICAL ANALYSIS | 25 |
| | 7.1 | DATA HANDLING RULES AND DEFINITIONS, INCLUDING HANDLING OF MISSING DATA | 25 |
| | 7.1 | SUBJECT DISPOSITION AND ANALYSIS POPULATIONS | |



Statistical Analysis Plan Protocol Nos.: PT010010 Date: 24 Aug 2017 

| | 7.3 | DEMOGE | RAPHIC AND BASELINE CHARACTERISTICS | 27 |
|---|---|---|---|---|
| | | 7.3.1 | Medical and Surgical History at Screening, Reproductive Status, and Pregnancy Te | |
| | | 7.3.2 | Prior and Concomitant Medications/Treatments | |
| | | 7.3.3 | Extent of Exposure to Study Medication and Compliance | 28 |
| | 7.4 | PHARMA | ACOKINETIC ASSESSMENTS | |
| | 7.5 | | Assessments | |
| | | 7.5.1 | Physical Examination | |
| | | 7.5.2 | Vital Signs | |
| | | 7.5.3 | 12-Lead Electrocardiogram | |
| | | 7.5.4 | Clinical Laboratory Tests | |
| | | 7.5.5 | Adverse Events | 33 |
| | | 7.5.6 | Urine Drug Screening and Alcohol Breath Testing | 33 |
| | | 7.5.7 | Pregnancy Test | |
| | | 7.5.8 | Prior/Concomitant Medications/Treatments | |
| 8. | ANA | LYSES I | PERFORMED BEFORE DATABASE CLOSURE | 34 |
| 9. | СНА | NGES F | ROM METHODS PLANNED IN THE PROTOCOL | 34 |
| 10. | STA | ΓISTICA | L SOFTWARE | 34 |
| 11. | REF | ERENCE | ES | 34 |
| APP | ENDI | X 1: DA | ΓA HANDLING RULES | 34 |
| APP | ENDI | X 2: TAI | BLE OF CONTENTS FOR END-OF-TEXT TABLES, LISTINGS, AND FIGU | RES.35 |
| A DD | ENDI | V 2. CT/ | CAE LABORATORY TEST CRITERIA FOR SHIFT TABLES AND CENTRA | A T |
| AFF | | | ORY REFERENCE RANGES FOR USE IN FLAGGING ABNORMAL VALUE | |



Statistical Analysis Plan Protocol Nos.: PT010010 Date: 24 Aug 2017 

#### **List of Tables**

| | Elist of Tubles | |
|---|---|---|
| Table 1 | Potentially Clinically Significant Criteria for Systolic and Diastolic Blood<br>Pressure Parameters | 20 |
| Table 2 | Potentially Clinically Significant Criteria for Heart Rate Parameters | 20 |
| Table 3 | List of Laboratory Tests | |
| Table 4 | Potentially Clinically Significant (PCS) Laboratory Parameter Criteria | 22 |
| | List of Figures | |
| Figure 1 | Study Design | 14 |





Protocol Nos.: PT010010 Date: 24 Aug 2017


#### LIST OF ABBREVIATIONS AND DEFINITIONS OF TERMS

AE Adverse event

ATC Anatomic Therapeutic Class

 $AUC_{0-12}$  Area under the plasma concentration-time curve from 0 to 12 hours

Auc<sub>0-t</sub> Area under the plasma concentration-time curve from 0 to the Time of the

Last Measurable Plasma Concentration

Au $C_{0-\infty}$  Area under the plasma concentration-time curve from 0 Extrapolated to

Infinity

BGF MDI Budesonide, Glycopyrronium, and Formoterol Fumarate Metered Dose

Inhaler

BID Bis in die, twice daily

BLOQ Below Limit of Quantification

BP Blood Pressure

CL/F Apparent Total Body Clearance

C<sub>max</sub> Maximum Plasma Concentration

COPD Chronic Obstructive Pulmonary Disease

ECG Electrocardiogram

EDTA Ethylenediaminetetraacetic Acid

eCRF Electronic Case Report Form

eg Exempli gratia; for example

FSH Follicle Stimulating Hormone

GFF MDI Glycopyrronium and Formoterol Fumarate Metered Dose Inhaler

GFR Glomerular Filtration Rate

HbsAg Hepatitis B Surface Antigen

hCG Human chorionic gonadotropin

HIV Human Immunodeficiency Virus

HR Heart Rate

IB Investigators Brochure



Protocol Nos.: PT010010
Date: 24 Aug 2017


ICF Informed Consent Form

i.e. Id Est; That Is

Pearl

IEC Independent Ethics Committee

IRB Institutional Review Board

 $\lambda_z$  Apparent Terminal Elimination Rate Constant

LLQ Lower Limit of Quantification

MDI Metered dose inhaler

MDRD Modification of Diet in Renal Disease

MedDRA Medical Dictionary for Regulatory Activities

μg Microgram mL Milliliter

mm Millimeter

mmHg Millimeter of mercury

msec (ms) Millisecond

NCA Non-Compartmental Analysis

PCS Potentially Clinically Significant

PFT Pulmonary Function Test

PK Pharmacokinetics

PR Pulse Rate

PT Preferred Term

PT003 Glycopyrronium and Formoterol Fumarate Inhalation Aerosol

PT010 Budesonide, Glycopyrronium, and Formoterol Fumarate Inhalation

Aerosol

QTcF QT Corrected Using Fridericia's Formula

 $RAC(C_{max})$  Accumulation ratio for  $C_{max}$ 

RAC(AUC<sub>0-12</sub>) Accumulation ratio for AUC<sub>0-12</sub>

SAE Serious adverse event

SAP Statistical Analysis Plan



**Statistical Analysis Plan** 

Protocol Nos.: PT010010 Date: 24 Aug 2017 

SOC System Organ Class

SOP Standard Operating Procedure

 $t_{1/2}$  Apparent Terminal Elimination Half-life

TEAE Treatment-emergent adverse event

TFL Table, Figure, Listing

 $t_{max} \hspace{1.5cm} Time \hspace{0.1cm} To \hspace{0.1cm} Maximum \hspace{0.1cm} Plasma \hspace{0.1cm} Concentration$ 

Vd/F Apparent Volume of Distribution

WHO World Health Organization



Statistical Analysis Plan Protocol Nos.: PT010010 Date: 24 Aug 2017 

## Trademark Information

| Trademarks Not Owned By Pearl |
|-------------------------------|
| Oxis |
| Pulmicort |
| Respules |
| Spiriva |
| Symbicort |
| Turbuhaler |
| Vacutainer |
| Ziploc |



Protocol Nos.: PT010010 Date: 24 Aug 2017 

#### 1. INTRODUCTION

This Statistical Analysis Plan (SAP) outlines the statistical methods for the display, summary and analysis of data to be performed at the end of Pearl Therapeutics, Inc. (Pearl) Study PT010010. The SAP should be read in conjunction with the study protocol and the electronic Case Report Forms (eCRFs) for the study. This version of the SAP has been developed using the PT010010-03 Amended Protocol (Version 4.0 dated 12 May 2017) and the CRF Revision 2 dated 2 March, 2017. This is the main SAP, describing the statistical analyses that will be carried out at the end of the study.

This is a phase I, randomized, double-blind, parallel-group, study to assess the pharmacokinetics (PK) and safety of two dosage strengths of PT010 (BGF MDI 320/14.4/9.6  $\mu$ g ex-actuator and (BGF MDI 160/14.4/9.6  $\mu$ g ex-actuator) and a single dosage strength of PT003 (GFF MDI 14.4/9.6  $\mu$ g ex-actuator) in healthy Chinese adult subjects following a single administration and after chronic administration for 7 days.

The definitions of data sets will be described in separate documents called SDTM specifications and ADaM specifications. A prototype SAS code appendix will not be necessary for this study because the statistics are descriptive in nature, without modeling or hypothesis testing.

#### 2. STUDY OBJECTIVES AND ENDPOINTS

#### 2.1 Study Objectives

#### 2.1.1 Primary Objective

• To assess the pharmacokinetic profile of two dosage strengths of BGF MDI (BGF MDI 320/14.4/9.6 µg ex-actuator and (BGF MDI 160/14.4/9.6 µg ex-actuator) and a single dosage strength of GFF MDI (GFF MDI 14.4/9.6 µg ex-actuator) in healthy Chinese adult subjects after a single administration and after chronic administration for 7 days.

#### 2.1.2 Secondary Objective

• To assess the safety and tolerability of two dosage strengths of BGF MDI and a single dosage strength of GFF MDI in healthy Chinese adult subjects after single administration and after chronic administration for 7 days.

#### 2.2 Study Endpoints

#### 2.2.1 Pharmacokinetic Endpoint

Pharmacokinetics of BGF MDI and GFF MDI will be assessed and compared using plasma concentrations of budesonide, glycopyrronium, and formoterol. For the single dose administration, time points for PK blood sample collection will be pre-dose within 60 minutes and post-dose at 2, 6, 20, and 40 minutes and at 1, 2, 4, 8, 10, 12, and 24 hours. Following 7 days

Protocol Nos.: PT010010 Date: 24 Aug 2017


of chronic dosing BID, time points for PK blood sample collection will be pre-dose within 60 minutes and post-dose at 2, 6, 20, and 40 minutes and at 1, 2, 4, 8, 10, 12 and 24 hours.

Pharmacokinetic parameters calculated at the first day (Day 1) and last dose (Day 8) during the Treatment Period will include the following:

- Maximum plasma concentration (C<sub>max</sub>)
- Area under the plasma concentration-time curve from 0 to 12 hours (AUC<sub>0-12</sub>)
- Time to maximum plasma concentration (t<sub>max</sub>)

The following PK parameters will be calculated at Day 1 only:

- Area under the plasma concentration-time curve from 0 to the time of the last measureable plasma concentration ( $AUC_{0-t}$ )
- Area under the plasma concentration-time curve from 0 extrapolated to infinity (AUC<sub>0- $\infty$ </sub>)
- Elimination half-life (t<sub>1/2</sub>)
- Apparent total body clearance (CL/F)
- Apparent volume of distribution (Vd/F)
- Apparent terminal elimination rate constant  $(\lambda_z)$

The following will be derived by taking subject level ratios of Day 8 values to Day 1 values:

- Accumulation ratio for C<sub>max</sub> (RAC [C<sub>max</sub>])
- Accumulation ratio for AUC<sub>0-12</sub> (RAC [AUC<sub>0-12</sub>])

#### 2.2.2 Secondary Endpoint

The safety and tolerability of BGF MDI and GFF MDI will be assessed from physical examination findings, AE (adverse event) reporting including serious adverse event (SAE) reporting, vital signs (blood pressure [BP], pulse rate [PR], respiratory rate, and body temperature), clinical laboratory values (hematology, chemistry, and urinalysis), and findings from 12-lead safety electrocardiograms (ECG) incorporated in the adverse events tabulation.

#### 3. STUDY DESIGN AND ANALYTICAL CONSIDERATIONS

#### 3.1 Study Design

This is a Phase I, single-center, randomized, double-blind, parallel-group, study to assess the PK and safety and tolerability of two doses of BGF MDI and a single dose of GFF MDI in healthy

Protocol Nos.: PT010010 Date: 24 Aug 2017 

Chinese adult subjects. Pharmacokinetics will be assessed following a single administration and after chronic administration for 7 days. Safety will be assessed during the 8-day treatment period and throughout the entire study until subjects are released from participation. All study drugs will be administered by oral inhalation. It is planned that the study will enroll and randomize an estimated 96 eligible subjects to one of three treatment groups in a 1:1:1 ratio to have approximately 90 completed subjects. Subjects will receive one of the following three treatments:

BGF MDI 320/14.4/9.6 μg

BGF MDI 160/14.4/9.6 μg

GFF MDI 14.4/9.6 μg

This study includes a Screening Period of up to 28 days and a single Treatment Period of 8 days. A follow-up phone call will be conducted at least 5 days, but no longer than 7 days after completion of the last dose. The maximum participation in the study for each subject is not expected to exceed approximately 43 days.

#### 3.1.1 Overall Study Design and Plan

The overall study design is summarized and illustrated in Figure 1.

Figure 1 Study Design



<sup>&</sup>lt;sup>\*</sup>24 hour PK following s single administration on Day 1

**Note**: All study drugs are administered by oral inhalation. A single dose of study drug will be administered on Day 1 and BID doses will be administered Day 2 through Day 7 of the Treatment Period, with a final single administration of study drug occurring on the morning of Day 8. Administration of study drug should occur at approximately the same time of day.

<sup>&</sup>lt;sup>1</sup>24 hour PK on Day 8 following a final single dose after twice daily chronic administration for 7 days





Protocol Nos.: PT010010 Date: 24 Aug 2017 

Subjects who provide informed consent, undergo Screening procedures, and qualify for the study will be randomized in a 1:1:1 ratio to one of three treatments: BGF MDI ( $320/14.4/9.6~\mu g$ ), BGF MDI ( $160/14.4/9.6~\mu g$ ), or GFF MDI ( $14.4/9.6~\mu g$ ). Approximately 32 subjects will be randomized to each treatment arm.

Subjects will be admitted as inpatients to the Clinical Research Unit (hereinafter referred to as "clinic") during the Treatment Period. For the Treatment Period, subjects will be admitted to the clinic on Visit 2 (the day prior to dosing), at which time, continuing eligibility will be assessed. At in-clinic Visit 3 (Day 1 of Treatment), if the subject continues to meet eligibility criteria, the subject will be randomized into the study, admitted into the inpatient study unit and administered their first single dose of study drug.

During the inpatient treatment period, study specified procedures will be performed and will include safety assessments, baseline and pre-, post-dose serial blood draws as defined in Protocol Section 7.3 and in Table 8—1, 8—2, and Table 8—3 of the study protocol. After all protocol specified assessments are completed and safety data has been reviewed by the Principal Investigator (Investigator) or designated staff, the subjects will be discharged from the clinic on Day 9. A follow-up phone call will be conducted 5 days, but no later than 7 days, after the last dose on Day 8.

# 3.1.2 Prior, Concomitant, Post-Treatment, Prohibited Medications, and Other Restrictions

Investigational therapies are not permitted within 30 days or five half-lives (whichever is longer) prior to beginning the Screening Period.

The use of prescription or over-the counter medications are not permitted within 30 days or five half-lives (whichever is longer) prior to Visit 3 (Day 1).

Acetaminophen will be permitted at doses of  $\leq 2$  grams/day as determined to be necessary by the Investigator or medically qualified designee.

With the exception of, contraceptives in female subjects, or need for medication during an emergency ongoing treatment for chronic conditions will not be allowed. Any medications that were being taken prior to signing the informed consent form (ICF) will be documented as prior study drugs and must be stopped prior to entry.

#### 3.1.2.1 Surgical Procedure/Intervention Restrictions

Major surgical interventions are not permitted within 4 weeks of study drug administration (Visit 3) and minor surgical interventions are not allowed within 2 weeks of study drug administration (Visit 3).

Protocol Nos.: PT010010 Date: 24 Aug 2017 

#### 3.1.2.2 **Dietary Restrictions**

Fasting (at least 8 hours) is required for scheduled complete clinical laboratory testing – chemistry and hematology (including glucose and potassium), at Screening Visit 1, Visit 2 (Day -1) and for the 24 hours post-dose sample collection on Day 9.

Fasting is not required for glucose and potassium only blood sample collections on Visit 3 (Day 1) at 30 min and at 2 hours post-dose and on Visit 4 (Day 8) at 30 min, 2 hours and 12 hours post-dose.

Standardized meals will be administered at specified times after observation of fasting time for blood draws. There are no restrictions regarding clear fluid intake.

Subjects are not allowed to consume grapefruits or grapefruit juice throughout the study. Subjects must not ingest xanthine (caffeine)-containing foods, beverages or medications for at least 6 hours prior to each study visit and for the duration of each study visit. Examples of such products include coffee, tea, chocolate, and cola. Decaffeinated beverages are acceptable.

#### 3.1.2.3 Illicit Drugs and/or Drugs of Abuse Restriction

Illicit drugs and/or drugs of abuse will not be allowed from within 1 year of Screening to whenever the subject discontinues the study. If any illicit drugs or drugs of abuse are used by the subject during the study, the dates of use and the amount will be documented.

#### 3.1.2.4 Smoking Restrictions

Smoking is prohibited throughout the duration of the study and 3 months prior to screening. Electronic cigarettes and nicotine supplements will be treated the same way as smoking is considered in the protocol.

#### 3.2 Randomization and Blinding

Following determination of study eligibility, subjects will be randomized in a 1:1:1 ratio to one of the three treatment groups: BGF 320/14.4/9.6  $\mu$ g, BGF 160/14.4/9.6  $\mu$ g, or GFF MDI 14.4/9.6  $\mu$ g.

All treatment arms will be double-blinded.

Randomization numbers will be generated off-site, to ensure allocation concealment, using a permutated block randomization design. The randomization numbers will be printed on sealed envelopes and corresponding component ID codes will be provided within the envelopes. The sealed envelopes are given out sequentially (i.e. there are serially numbered opaque sealed envelopes). Sealed emergency unblinding envelopes will also be provided separately.

Subjects, investigators and the sponsor will be blinded to the treatment administered as described above until the study database is locked. The pharmacist will have access to the unblinded randomized treatment sequence.





Protocol Nos.: PT010010 Date: 24 Aug 2017 

#### 3.3 Hypothesis Testing

No formal hypothesis tests will be performed for this study.

#### 3.4 Interim Analysis

There is no interim analysis planned for this study.

#### 3.5 Sample Size

| Previous studies with BGF MDI suggest that | the inter-subj | ect variability | of glycopyr | ronium after | r |
|---|---|---|---|---|---|
| single-dose administration may be as high as | | | | | |

#### 3.6 Study Procedures

Study procedures are contained in Table 8—1, 8—2, and Table 8—3 of the study protocol.

#### 3.7 Schedule of Assessments

A schedule of events is provided in Table 8—1 of the study protocol. Detailed schedules of inpatient assessments on Visit 3 (Day 1) and Visit 4 (Day 8) are provided in Table 8—2 and Table 8—3, respectively, of the study protocol.

#### 4. DATA AND ANALYTICAL QUALITY ASSURANCE

The overall quality assurance (QA) procedures for the study data, statistical programming and analyses are described in Standard Operating Procedures (SOPs) of Detailed data management procedures are documented in the study Data Management Plan, and Data Validation Check Specifications, and Integrated Safety Data Review Plan. Detailed statistical and programming quality control and quality assurance procedures are documented in the Statistical Analysis and Programming QC/QA Plan.

The study endpoints and analytic approaches are both prospectively defined and documented in the protocol and in this SAP. The SAP will be finalized, and protocol violations will be identified and decisions for inclusion and exclusion of subjects from the PK Population will be made at the Blinded Data Review Meeting (BDRM) prior to the database lock and data analysis.

#### 5. ANALYSIS POPULATIONS

#### **5.1** Population Definitions

## 5.1.1 Safety Population

The **Safety Population** is defined as all subjects who receive at least one dose of any blinded study drug.

Protocol Nos.: PT010010 Date: 24 Aug 2017 

Safety analyses will be performed on data from all subjects in the Safety Population. Analyses will be according to treatment received.

#### 5.1.2 Pharmacokinetic (PK) Population

The **PK Population** is defined as all subjects in the Safety Population who have sufficient data to reliably calculate at least one PK parameter and do not have major protocol deviations (to be determined at the BDRM prior to unblinding). A major protocol deviation is a protocol deviation which can affect membership in an analysis population.

Pharmacokinetic analyses will be performed on data from all subjects in the PK Population. Analyses will be according to treatment received.

#### **5.2** Populations for Analyses

Demographics and baseline characteristics will be summarized descriptively for the PK and Safety Populations. Extent of exposure will also be summarized for the Safety and PK Populations. For the PK Population, descriptive statistics without model adjustment will be used to describe the budesonide, glycopyrrolate and formoterol PK parameters after treatment with two dosage strengths of BGF MDI and single dosage strength of GFF MDI. The Safety Population will be used to summarize safety. Safety and tolerability analyses will be based on descriptive statistics for vital signs, physical examination and laboratory measurements as appropriate, and also on frequencies of AEs (including any AEs based on ECG findings) as well as the number and proportion of subjects with AEs.

#### 6. SPECIFICATION OF ENDPOINTS AND VARIABLES

#### 6.1 Demographics and Baseline Characteristics

General demographic information such as age, race/ethnicity, gender, weight, and height will be collected at the Screening visit. Age will be calculated as the integer part of (Informed Consent date – Birth date)/365.25.

Medical/surgical history will be collected on the eCRF during the Screening period. Medical history will be coded using the latest version of the Medical Dictionary for Regulatory Activities (currently MedDRA 19.1). Serology testing for HIV, HBsAg, Syphilis Ab, and Hepatitis C antibody will be conducted at the Screening visit.

The definitions for the derived demographic or baseline characteristic variables can be found in Appendix 1.

#### 6.2 Pharmacokinetics

See Section 7.4.

Protocol Nos.: PT010010 Date: 24 Aug 2017 

#### **6.3** Safety Assessments

## 6.3.1 Physical Examination

Any clinically significant physical examination abnormality reported after the start of study medication will be reported as an adverse event. These adverse events will be included in the AE summaries.

The physical examination will include:

- Documentation of height (Screening only)
- Documentation of weight (Screening only)
- General appearance
- Head, eyes, ears, nose, and throat
- Respiratory
- Cardiovascular
- Musculoskeletal
- Abdominal
- Neurologic
- Extremities
- Dermatologic
- Lymph nodes

#### 6.3.2 Vital Signs

Vital sign determinations, including BP, PR, respiratory rate, and body temperature will be performed after the subject has been supine for a 5-minute period at the Screening Visit, on the day of clinic admission Visit 2 (Day -1), Days 2 through Day 7, and on Visit 3 (Day 1) and Visit 4 (Day 8) within 120 minutes (on Day 1; within 60 minutes on Day 3) prior to administration of study drug and 30 minutes, 2 hours, 4 hours, 12 hours, and 24 hours post administration of study drug.

Potentially clinically significant (PCS) changes in systolic and diastolic blood pressure will be defined based on the following criteria provided by Pearl, Inc.:

Protocol Nos.: PT010010 Date: 24 Aug 2017 

Table 1 Potentially Clinically Significant Criteria for Systolic and Diastolic Blood Pressure Parameters

| Parameter (mmHg) | Post-Baseline Criteria |
|------------------------------------|--------------------------------|
| Systolic Blood Pressure, increase | ≥180 mmHg and increase from |
| | baseline ≥20 mmHg |
| Systolic Blood Pressure, decrease | ≤90 mmHg and ≥20 mmHg decrease |
| | from baseline |
| Diastolic Blood Pressure, increase | ≥105 mmHg and increase from |
| | baseline ≥15 mmHg |
| Diastolic Blood Pressure, decrease | ≤50 mmHg and ≥15 mmHg decrease |
| | from baseline |

Potentially clinically significant (PCS) changes in heart rate will be assessed as follows:

 Table 2
 Potentially Clinically Significant Criteria for Heart Rate Parameters

| Parameter | Post-Baseline Criteria |
|-------------------|------------------------------------------|
| Tachycardia Event | ≥110 bpm and increase ≥15% from baseline |
| Bradycardia Event | ≤50 bpm and decrease ≥15% from baseline |

#### 6.3.3 12-Lead Electrocardiogram

Any clinically significant abnormality noted post-randomization based on twelve-lead safety ECGs will be recorded as adverse events.

Machine-read ECG parameter data will be provided to the Investigator by local ECG lab(s).

#### **6.3.4** Clinical Laboratory Tests

Laboratory testing (hematology with differential, chemistry and urinalysis) will be performed using standard methods.

Standardized meals will be administered at specified times after observing fasting times for blood draws.

Potentially Clinically Significant Laboratory Values Above/Below a Clinically Relevant Threshold on-treatment, based on CTCAE 4.03 and other criteria, will be identified based on the thresholds in Table 4.

Protocol Nos.: PT010010 Date: 24 Aug 2017 

**Table 3** List of Laboratory Tests

| Hematology | Blood Chemistry | |
|---|---|---|
| Hematocrit <sup>a</sup> | Creatinine <sup>b</sup> | Bilirubin (direct) |
| Hemoglobin | Potassium (K+) <sup>c</sup> | Alanine aminotransferase |
| Serum Iron | Sodium (Na+) | (ALT) |
| Ferritin | Chloride (Cl-) | Aspartate aminotransferase (AST) |
| Platelet count | Magnesium (Mg++) | Gamma- |
| Red blood cell (RBC) count | Calcium | Glutamyltransferase |
| White blood cell (WBC) count | Inorganic phosphate | (GGT) |
| WBC differential | Glucose <sup>c</sup> | Alkaline phosphatase |
| Mean corpuscular volume (MCV) | Uric Acid | Total Protein |
| Mean cell haemoglobin (MCH) | Bilirubin (Total) | Albumin |
| MCH concentration (MCHC) | Blood Urea Nitrogen (BUN) | Albullilli |

**Urinalysis:** Macroscopic examination routinely including specific gravity, pH, protein, glucose, ketones, blood and urobilinogen. A microscopic examination will be performed if warranted based on macroscopic results.

**Urine drug screen:** A urine sample will be collected and analyzed (positive or negative) for drugs of abuse including amphetamine, opiate, cocaine, barbiturates, benzodiazepines, and marijuana [tetrahydrocannabinol (THC)].

**Breathalyzer Test:** A breathalyzer test will be performed for the presence of alcohol (positive or negative).

**Serology:** Testing for HbsAg, Hepatitis C antibody and HIV will be performed at screening only. Results of each serology test will be reported as either positive or negative.

For females who are not post-menopausal: A <u>serum hCG</u> test at the screening visit and <u>urine hCG</u> test at admission.

For females of non-childbearing potential: A <u>serum hCG</u> test at the screening visit and <u>urine hCG</u> test at admission. In addition, a serum, follicle-stimulating hormone (FSH) test for confirmation of non-childbearing status will be performed at screening only.

Abbreviations: eGFR=estimated glomerular filtration rate; HbsAg=hepatitis B surface antigen; hCG=human chorionic gonadotropin; HIV=human immunodeficiency virus; FSH=follicle-stimulating hormone.

#### C-MDRD (modified for Chinese) equation:

eGFR =  $175 \times (Serum Creatinine) - 1.234 \times (Age) - 0.179 \times (0.79 \text{ if Female})$ 

<sup>&</sup>lt;sup>a</sup> Packed cell volume (PCV).

<sup>&</sup>lt;sup>b</sup> eGFR will be calculated by the Modification of Diet in Renal Disease (MDRD) equation following : http://www.columbiamedicine.org/divisions/gharavi/calc\_egfr.php

<sup>&</sup>lt;sup>c</sup> Additionally, within 60 minutes prior to dosing and at 30 min, 2 hours, and 12 hours (Visit 4 only) post-dose of Treatment.

Protocol Nos.: PT010010 Date: 24 Aug 2017 

#### Table 4 Potentially Clinically Significant (PCS) Laboratory Parameter Criteria

| Parameter | Post-Baseline Criteria |
|--------------------------------|------------------------------------------|
| Hematology | |
| Hemoglobin | <8.0 g/dL (<80 g/L) |
| | Increase of >40 g/L to a value above the |
| | ULN |
| White Blood Cell Count | $<2000/\mu$ L |
| | >35,000/μL |
| Platelet Count | <50,000/μL |
| | >999,000/μL |
| Chemistry | |
| eGFR-EPI | <30 mL/min/1.73 m <sup>2</sup> |
| AST | >3 x ULN |
| ALT | >3 x ULN |
| Alkaline Phosphatase | >5 x ULN |
| Total Bilirubin | >2 x ULN |
| Blood Glucose* (random values) | <2.2 mmol/L (<39.6 mg/dL) |
| | >13.9 mmol/L (>250 mg/dL) if baseline |
| | is below 10.0 mmol/L (180 mg/dL), > |
| | 16.7 mmol/L (>300 mg/dL) if baseline |
| | is greater than 10.0 mmol/L (180 |
| | mg/dL) |
| Serum Potassium | <3.0 mmol/L |
| | >6.0 mmol/L |

<sup>\*</sup>CTCAE 4.03 criteria are based on fasting glucose values. However, subjects were not required to fast prior to obtaining blood glucose values.

#### **6.3.5** Adverse Events

Adverse events (AEs) will be collected from the time of administration of the first dose of study drug to the time of the Follow-Up Telephone Call Visit, study termination, or study exit. AEs will be characterized by severity and relationship to study drug. The incidence of an adverse event will be defined by the number of subjects experiencing an event.

Adverse events will be collected and coded using the latest version of MedDRA available at the time of database lock for this study. The study physician will review the adverse event coding.

Adverse events that occur between the time the subject signs the informed consent form for the study and the time when that subject is randomized will be summarized as medical history and not as a treatment-emergent adverse event (TEAE).





Protocol Nos.: PT010010 Date: 24 Aug 2017 

An AE is considered treatment-emergent (TEAE) if the date of onset is on or after the date of first dose of study drug in the study until the final Telephone Follow-up. Adverse events will be listed in adverse event data listings (*Listing 7.1*).

**Events with Irregular Start Dates**: All adverse events will be included in the tabulations regardless of the completeness of the onset dates.

Adverse events include, but are not limited to:

- Any symptom or condition not previously reported by the subject (medical history).
- An exacerbation of a pre-existing symptom or condition.
- A significant increase in frequency or intensity of a pre-existing episodic event or condition.
- A drug interaction.
- A condition first detected or diagnosed after study drug administration even though it may have been present prior to the start of the study.
- Medical or surgical procedures (e.g., surgery, endoscopy, tooth extraction, blood transfusion) are not considered AEs and the condition that results in the procedure is considered an AE (e.g., bleeding esophageal varices, dental caries).

#### An AE does **not** include:

- Overdose of either study drug or concurrent medication without any clinical signs or symptoms.
- Non-clinically significant abnormal laboratory values. (If accompanied by signs/symptoms, the signs or symptoms are considered an AE).

An AE is considered "serious" if, in the view of the Investigator or Sponsor, it results in any of the following outcomes:

- Death
- A life-threatening AE
- In patient hospitalization or prolongation of existing hospitalization





Protocol Nos.: PT010010 Date: 24 Aug 2017 

- A persistent or significant incapacity or substantial disruption of the ability to conduct normal life functions
- A congenital anomaly/birth defect.

Important medical events that may not result in death, be life threatening, or require hospitalization may be considered serious when, based upon appropriate judgment, they may jeopardize the subject and may require medical or surgical intervention to prevent one of the outcomes listed in the definition. Examples of such medical events include allergic bronchospasm requiring intensive treatment in an emergency room or at home, blood dyscrasias or convulsions that do not result in subject hospitalization, or the development of drug dependency or drug abuse.

Hospitalization for a pre-existing condition, including elective procedures, which has not worsened, does not constitute an SAE.

An AE is considered "life-threatening" if, in the view of the Investigator or Sponsor, its occurrence places the subject at immediate risk of death. It does not include an adverse reaction or suspected adverse reaction that, had it occurred in a more severe form, might have caused death.

An unexpected AE means any AE in which the specificity or severity is not consistent with the current Investigator's Brochure (IB).

Many laboratory abnormalities observed during the course of a study will be included under a reported AE describing a clinical syndrome (e.g., elevated BUN and creatinine in the setting of an AE of renal failure, or decreased hemoglobin in a case of bleeding esophageal varices). In such cases, the laboratory abnormality itself (e.g., elevated creatinine in a setting of renal failure) does not need to be recorded as an AE. However, isolated laboratory abnormalities should be reported as AEs if they are considered to be clinically significant by the Investigator.

Criteria for a "clinically significant" laboratory abnormality are:

- A laboratory abnormality that leads to a dose-limiting toxicity (e.g., an abnormality that results in study drug dose reduction, suspension, or discontinuation)
- A laboratory abnormality that results in any therapeutic intervention (e.g., concomitant medication or therapy)
- Other laboratory abnormality judged by the Investigator to be of any particular clinical concern (e.g., significant fall in hemoglobin not requiring transfusion)

Protocol Nos.: PT010010 Date: 24 Aug 2017 

For laboratory abnormalities that do not meet the above criteria but are outside of normal range (e.g., < or > normal reference range), the Investigator should indicate whether the value is potentially clinically significant (Table 4) or not clinically significant for the subject.

#### 6.3.6 Urine Drug Screening/Alcohol Breath Testing

A urine sample will be collected and analyzed (positive or negative) for drugs of abuse including amphetamine, opiate, cocaine, barbiturates, benzodiazepines, and marijuana [tetrahydrocannabinol (THC)]. A breathalyzer test will be performed for the presence of alcohol (positive or negative). Both tests will be conducted at the Screening Visits 1 and 2.

#### 6.3.7 Pregnancy Test

A serum hCG test and a urine hCG test at the Screening visit will be conducted for all females.

#### **6.3.8** Concomitant Medications/Treatments

Concomitant medications will be collected for all visits of the study.

Any medications that were being taken prior to signing the ICF will be documented as prior study medications and must be stopped prior to entry.

Concomitant medications will be coded using the latest version of the World Health Organization (WHO) Drug Dictionary Enhanced (WHO DDE) and the WHO Herbal Dictionary (WHO-HD).

#### 7. STATISTICAL ANALYSIS

All data collected on the CRF and contributing to the analysis will be provided in listings, except for data collected only for confirmation of study entry criteria and for study management purposes. Data for all subjects who are randomized will be included in the subject data listings. Data for non-randomized subjects will be listed where available.

All PK and safety parameters will be summarized by treatment unless specified otherwise.

Continuous variables will be summarized with descriptive statistics: the number of non-missing values, mean, standard deviation, median, minimum, and maximum.

Categorical variables will be summarized with frequency counts and percentages (where appropriate).

#### 7.1 Data Handling Rules and Definitions, Including Handling of Missing Data

Missing data will be maintained as missing in the analysis datasets, unless specified otherwise. For variables where missing data are imputed, the analysis dataset will contain a new variable with the imputed value, and the original variable value will be maintained as missing.





Protocol Nos.: PT010010 Date: 24 Aug 2017 

#### Data Imputation for Pharmacokinetic Summaries

Data imputation for pharmacokinetic summaries is detailed in Section 7.4.

#### Data Imputation for Adverse Events Summaries by Severity and Relationship to Study Drug

For the AE summaries by severity, an AE with missing severity will be deemed as severe. For AEs that could be associated with any study procedure the causal relationship is implied as 'yes'. Imputed values will not be listed in data listings.

#### Data Imputation for Laboratory, Vital Sign, and ECG Summaries (Continuous Parameters)

By-visit and by-timepoint summaries will be based on scheduled visits and/or timepoints (i.e. no time windows), as applicable. Data from unscheduled visits and/or timepoints will not be used for by-visit or by-timepoint summaries but will be included in the listings. Data from both scheduled and unscheduled visits will be used for the end-of-treatment summary, for shift tables and for determining incidence of clinically significant values. End-of-treatment refers to the last visit during study treatment when an assessment was made.

#### Data Imputation (All Laboratory Summaries)

Laboratory values of '>=x' or '<=x' will be taken as the value of x in the analyses. If a laboratory value is prefixed with'>': the available original value +0.001 will be used for table summaries; if a laboratory value is prefixed with '<', then the original value -0.001 will be used in table summaries.

#### Study Dates and Day of Assessment or Event

Study Day and Day of Assessment or Event definitions are provided in Appendix 1, Data Handling Rules.

#### 7.2 Subject Disposition and Analysis Populations

A disposition table for all subjects screened will be provided (*Table 1.1*). A flow chart of subject distribution will also be provided (*Figure 1.1*). This tabulation will include the number and percentage of subjects in each randomized treatment who were treated with the study treatment, who discontinued treatment prematurely, who withdrew from the study prematurely, and who completed the study. The number and percentage of randomized subjects included in the Safety and PK Populations will also be tabulated (*Table 1.3*). Informed consent is listed in *Listing 1.1*.

A summary of reasons for withdrawal from study treatment will be summarized for the Safety Population (*Table 1.2*). These reasons will be listed in *Listing 1.2*.



Protocol Nos.: PT010010 Date: 24 Aug 2017 

#### 7.3 Demographic and Baseline Characteristics

Demographic data will be summarized by treatment group for both the Safety and PK Populations (Tables 1.4.1 and 1.4.2). Continuous demographic and baseline variables will be summarized by tabulating the number of subjects, mean, standard deviation (SD), median, minimum, and maximum values in each treatment group. For categorical demographic and baseline variables, the frequency and percentage of subjects in each treatment group will be tabulated. Demographic data will be listed (Listing 1.1). Baseline information (including Serology Testing (Listing 4.1) and Medical and Surgical History (Listing 4.2)) will be listed.

Demographic variables summarized will include the following:

- Age
- Gender
- Race
- Ethnicity
- Smoking Status (including number of years smoked, time in years since last smoked)
- Weight
- Height
- BMI (body mass index, derived from weight and height, equal to weight in kg divided by the square of height in m)

# 7.3.1 Medical and Surgical History at Screening, Reproductive Status, and Pregnancy Testing

Relevant medical history, based on the opinion of the Investigator, will be obtained from the subject at Screening, and recorded on the source document. Medical history will capture the subject's family health history, history of hospitalization, and history of surgeries.

Medical and Surgical History at Screening will be listed for all randomized subjects (*Listing 4.2*).

Screening Reproductive Status and Pregnancy Testing Results will be listed (*Listing 10.4*).

#### 7.3.2 Prior and Concomitant Medications/Treatments

**Coding:** Verbatim medication/treatment terms will be coded by will be assigned a preferred term and an ATC (anatomic therapeutic class) term using the latest version of the World Health Organization Drug Dictionary (WHO-DD) available (version: 3Q 2016 or later).

**Multiple ATC assignments:** If there are multiple ATC codes assigned to the same concomitant medication, the "primary" one based on medical evaluation by study physician will be used. All





Protocol Nos.: PT010010 Date: 24 Aug 2017 

prior medication taken by the subject within 30 days of Screening for the study and all concomitant therapy taken by the subject while on study will be recorded in the eCRF.

**Prior medication/treatment** is any medication/treatment taken prior to study treatment, even if this medication continued to be taken on the day of the start of study treatment in the study or afterward (*Appendix 1*).

Concomitant medication/treatment is any medication/treatment reported as being taken after the start of the study treatment in the study and being taken on or before the date prior to completion of or discontinuation from study treatment for the subject. A medication with an onset date on or after the date of discontinuation from or completion of randomized study treatment for the subject will not be considered concomitant, but will be considered a Post-Treatment medication/treatment.

Any medication/treatment which cannot be identified as Prior, Concomitant, or Post-Treatment will be considered as being in each of the categories that are possible from the available information.

Prior, concomitant, and post-treatment medications will be listed (Listing 10.1).

#### 7.3.3 Extent of Exposure to Study Medication and Compliance

Subject's exposure to a study treatment will be determined by the duration of time (days) for which the doses were administered, defined as "((End date of treatment – Date of first dose of treatment) + 1)". Percent compliance is defined as (total number of puffs of study treatment taken on a study day/total expected puffs taken on a study day) averaged across all days of a subject's dosing between start day of study treatment and last day on study treatment) x 100. For BGF MDI and GFF MDI, the expected number of puffs for a test day which is the last date of treatment will be 2, and the expected number of puffs for the last date of treatment which is not a test day will be 4 when a PM dose is taken but will be 2 otherwise; the expected number of puffs on dates prior to the last date of treatment will be 4.

The number of days of exposure to study treatment will be summarized for each treatment for the Safety Population. The tabulation will include the number and percentage of subjects with 1, 2, 3, 4, 5, 6, 7, and 8 days of exposure. The total person-years of exposure for a treatment group, defined as the total exposure in the study across all subjects in the treatment, will also be provided by treatment (*Table 1.6* for the Safety Population).

In addition, treatment compliance will be provided in this summary. The treatment compliance will be categorized into 7 different groups depending on the degree of compliance: 0 - <20%,  $\ge 20 - <40\%$ ,  $\ge 40 - <60\%$ ,  $\ge 60 - <80\%$ ,  $\ge 80 - \le 100\%$ ,  $>100 - \le 120\%$ , and >120%. Also provided in this summary will be descriptive statistics (n, mean, standard deviation, median, minimum and maximum) for percent compliance by treatment. Treatment compliance will be reported in *Listing 6*. A listing of treatment dosing and dispensing information will be provided





Protocol Nos.: PT010010 Date: 24 Aug 2017 

in *Listing 5*. Any comments related to study medication or any other additional study comments will be listed (*Listing 10.5*).

#### 7.4 Pharmacokinetic Assessments

For the single dose administration, time points for PK blood sample collection will be pre-dose within 60 minutes and post-dose at 2, 6, 20, and 40 minutes, and at 1, 2, 4, 8, 10, 12 and 24 hours.

Following 7 days of chronic dosing BID, time points for PK blood sample collection will be predose within 60 minutes and post-dose at 2, 6, 20, and 40 minutes, and at 1, 2, 4, 8, 10, 12 and 24 hours starting on the morning of the 8<sup>th</sup> day.

Actual sampling time points relative to dosing will be used for PK assessments and analysis where available. It is expected that the actual sampling time will generally be available. In any (likely rare) cases when the actual sampling time was not recorded, the scheduled time may be used. This is considered preferable to ignoring a valid concentration measurement.

The concentration-time data reported by the bioanalytical laboratory will be evaluated for inclusion in the PK analysis dataset.

The PK analysis will be performed for subjects in the PK Population.

PK parameters will be estimated by non-compartmental analysis (NCA) using the software

From the plasma budesonide, glycopyrronium and formoterol concentration-time data, the following PK parameters will be estimated for each subject where possible on Day 1 of the treatment period:

| $AUC_{0-t}$ | Area under the plasma concentration-time curve from 0 to the time of the last |
|---|---|
| | measurable plasma concentration |
| $AUC_{0-12}$ | Area under the plasma concentration-time curve from time 0 to 12 hours post dose |
| $\mathrm{AUC}_{0\text{-}\infty}$ | Area under the plasma concentration-time curve from time 0 extrapolated to |
| | infinity |
| $C_{max}$ | Maximum observed plasma concentration, expressed in concentration units |
| $t_{max}$ | Time to reach maximum observed plasma concentration (C <sub>max</sub> ), expressed in |
| | minutes |
| $\lambda_{\mathrm{z}}$ | Terminal elimination rate constant, calculated from the slope of the terminal |
| | portion of the ln(drug concentration) versus time curve |
| $t_{1/2}$ | Apparent terminal elimination half-life, expressed in hours, calculated as $\ln 2/\lambda_z$ |
| CL/F | Apparent total body clearance |
| Vd/F | Apparent volume of distribution |





Protocol Nos.: PT010010 Date: 24 Aug 2017 

From the plasma budesonide, glycopyrronium and formoterol concentration-time data, the following PK parameters will be estimated for each subject where possible on Day 8 during the treatment period:

| $AUC_{0-12}$ | Area under the plasma concentration-time curve from time 0 to 12 hours post dose |
|---|---|
| $C_{max}$ | Maximum observed plasma concentration, expressed in concentration units |
| t <sub>max</sub> | Time to reach maximum observed plasma concentration (C <sub>max</sub> ), expressed in hours |

 $AUC_{0-t}$ ,  $AUC_{0-12}$ , and  $AUC_{0-\infty}$ , will be calculated using the linear-log trapezoidal method.

The PK parameters  $C_{max}$  and time to  $C_{max}$  ( $t_{max}$ ) will be obtained from the observed values.

 $\lambda_z$  will be estimated for each subject where feasible by linear regression analysis, calculated from the slope of the terminal portion of the ln(drug concentration) versus time curve. Selection of data points to include in the estimation of  $\lambda_z$  for each subject for each treatment for each analyte will be based on the following criteria:

- All samples used should preferably fall in the log-linear elimination phase.
- At least 3 samples above lower limit of quantification (LLQ) should be used in the estimation.
- C<sub>max</sub> must not be used in the estimation.

In order for the selection to take place the adjusted r<sup>2</sup> value reported in must be above 0.7.

 $t_{1/2}$  will be calculated as  $ln2/\lambda_z$ .

For the purposes of parameter estimation, plasma concentration values below the LLQ will be set to missing in the NCA with the exception of those values reported at Day 1 pre-dose. Day 1 pre-dose concentrations that are below the limit of quantification (BLOQ) will be set to zero (per SOP) for the NCA. Concentrations measured after the Day 1 dose of study medication that are BLOQ will set to missing values (per SOP) for the NCA. Missing values (e.g., no blood sample collected, no value obtained at analysis) will be treated as missing and excluded from the NCA. If there are ≥2 consecutive missing concentration values, the estimation of PK parameters will be evaluated on a case-by-case basis.

For descriptive statistics for concentrations and for the concentration figures, all values below LLQ will be assigned a value of ½ LLQ except for Day 1 pre-dose which will be assigned a value of 0 (no geometric mean will be calculated for Day 1 pre-dose).

In addition to the above PK parameters to be calculated on Day 1 and Day 8, accumulation ratios for  $AUC_{0-12}$  (RAC [AUC<sub>0-12</sub>]) and  $C_{max}$  (RAC [C<sub>max</sub>]) will be calculated by taking subject level ratios of Day 8 values to Day 1 values.





Protocol Nos.: PT010010 Date: 24 Aug 2017 

All concentration-time data reported by the bioanalytical laboratory, for each analyte, for each treatment, will be listed for subjects in the PK Population (*Listing 8.1*). Actual sample collection times will be detailed in the listing along with the scheduled nominal sample collection times. In addition, all calculated PK parameters for each treatment for each analyte will be listed (*Listing 8.2*).

Descriptive statistics for plasma concentrations of budesonide, formoterol, and glycopyrronium, by treatment, visit and time point will be summarized. Descriptive statistics will include the number of observations (n), mean (CV%), SD, standard error (SE), median, minimum (min), maximum (max), geometric mean, and geometric coefficient of variation ( $Tables\ 2.1.1,\ 2.2.1,\ and\ 2.3.1$ ). The geometric coefficient of variation (of a statistic y) is calculated as GEOCV(y) (%) = 100\*sqrt[(exp[var(ln[y])])-1], where sqrt is the square root function and "var" is variance.

Descriptive statistics for PK parameters of budesonide, glycopyrronium, and formoterol, will be summarized by treatment and visit. Descriptive statistics will include the number of observations (n), mean (CV%), SD, median, min, max, geometric mean, and geometric coefficient of variation. For the PK parameter t<sub>max</sub>, only the number of observations (n), mean, median, minimum (min), and maximum (max) will be presented (*Tables 2.1.2, 2.2.2, and 2.3.2*).

The plasma concentration-time profiles for individual and mean plasma concentrations of budesonide, formoterol, and glycopyrronium, will be presented for each treatment and each visit on the linear/linear scale and on the linear/log-linear scale.

Mean and individual plots will be separate for each analyte. Nominal sampling time points relative to dosing will be used for all mean plots. Actual sampling time points will be used for all individual plots (mean plots in *Figures 2.1.1* through *2.3.2* and individual plots in *Figures 2.4.1* through *2.6.2*).

#### 7.5 Safety Assessments

Safety data will be summarized by treatment and listed. The safety of BGF MDI and GFF MDI will be assessed from physical examination findings, AE reporting including SAE reporting, vital signs (BP, PR, respiratory rate, and body temperature), clinical laboratory values (hematology, chemistry, and urinalysis), and findings from 12-lead ECGs. The incidence of AEs and SAEs will be tabulated by treatment. Summary statistics of assessed laboratory values will be tabulated by treatment.

#### 7.5.1 Physical Examination

Any clinically significant physical examination abnormality reported after the start of study medication was to be reported as an adverse event. Thus, these will be included in listings of adverse events and summarized in adverse event summaries.





Protocol Nos.: PT010010 Date: 24 Aug 2017 

#### 7.5.2 Vital Signs

Vital sign measurements (PR, BP, body temperature, and respiratory rate) as collected on eCRFs (see Section 6.3.2) during the study will be displayed in a vital sign listing, as well as weight and height (collected at the Screening visit) (*Listing 10.2*).

Summary statistics (n, mean, median, standard deviation, minimum and maximum) of pre-dose (in the respective period) and post-dose values (in the respective period) as well as changes from baseline values for systolic blood pressure, diastolic blood pressure and pulse rate will be tabulated by treatment group (*Table 3.4.1*). Baseline is defined (computationally) as the mean of all available pre-dose measurements taken on Day 1 prior to the start of dosing with study drug.

The percentage of subjects with potentially clinically significant values for vital signs at any time post-dose at a visit will be summarized by treatment based on the criteria in Table 1 and Table 2 (*Table 3.4.2*). They will also be listed (*Tables 3.4.3* and *3.4.4*).

#### 7.5.3 12-Lead Electrocardiogram

All clinically significant abnormalities after the first dosing through the treatment period until follow-up telephone will be reported as TEAEs and followed closely by the Investigator in order to assure the safety of the study subject.

### 7.5.4 Clinical Laboratory Tests

Summary statistics (n, mean, median, standard deviation, minimum, and maximum) of assessment values for laboratory testing (hematology with differential (*Table 3.3.1*), serum chemistry including estimated eGFR (*Table 3.3.2 and 3.3.3*) will be tabulated by treatment group at each time point and at each visit. Urinalysis results will be listed (*Listing 9.3*) and tabulated (*Table 3.3.5*). Changes from baseline will also be summarized by treatment group at 24 hours post-dose at Day 8 (Visit 4). Baseline is the last assessment during the screening period (e.g. Visit 2).

Individual clinical laboratory variables for hematology, serum chemistry including estimated eGFR and urinalysis will be provided in listings (*Listings 9.1 - 9.3*).

Glucose and potassium will also be collected within 30 minutes and 2 hours post-dose at Visit 3, and 60 minutes pre-dose, and 30 minutes, 2 hours, 12 hours, and 24 hours post-dose at Visit 4. The values as well as the changes from baseline for each visit and time point will be summarized by treatment (Table 3.3.4). Baseline is the last assessment prior to the first dose of study treatment. Glucose and potassium are also included into the complete laboratory assessment at Visit 2.

For glucose and potassium, the frequency and percentage of potentially clinically significant values will be summarized by treatment group, at each post-dose timepoint (*Table 3.3.4*). Potentially clinically significant values for serum potassium and blood glucose may be found in Table 4 (CTCAE Version 4.03). Potentially clinically significant laboratory values for potassium, glucose, and other laboratory parameters will be listed (*Tables 3.3.6, 3.3.7, and 3.3.8*).





Protocol Nos.: PT010010 Date: 24 Aug 2017 

Shifts from baseline to 24 hours post-dose at Visit 4 (Day 9), based on reference ranges (Low, Normal, High), will be presented by treatment group for hematology and serum chemistry (*Table 3.3.9*) and for urinalysis (*Table 3.3.10*). Baseline is the last assessment during the screening period (e.g. Visit 2) for all laboratory assessments.

Many laboratory abnormalities observed during the course of a study will be included under a reported AE describing a clinical syndrome (e.g., decreased hemoglobin in a case of bleeding esophageal varices). In such cases, the laboratory abnormality itself (e.g., elevated creatinine in a setting of renal failure) does not need to be recorded as an AE. However, isolated laboratory abnormalities should be reported as AEs if they are considered to be clinically significant by the investigator.

#### 7.5.5 Adverse Events

Treatment-emergent AEs (TEAEs) will be included in tabular format, for subjects who meet the criteria for the Safety Population. Listings for AEs will present all AEs in the database for all subjects (*Listings 7.1 and 7.2*). All AEs, whether treatment-emergent or not, will be included in the Listings.

Analysis endpoints for AEs include both the numbers of treatment-emergent AEs as observed by the investigational team or reported by the subject, and the numbers of subjects experiencing treatment-emergent adverse events. The incidence of a TEAE will be defined as the number of subjects experiencing an event.

An overall table of subjects with at least one TEAE will be summarized by treatment group, for subjects with AEs related to study treatment, with SAEs, with SAEs related to study treatment, with AEs leading to early discontinuation from study treatment, with SAEs leading to early withdrawal from study treatment, and with deaths (*Table 3.1.1*).

The frequency and percentage of subjects experiencing a specific AE will be tabulated by system organ class (SOC) and preferred term (PT) by treatment group for the Safety Population (*Table 3.1.2*).

TEAEs will be summarized by (maximum) severity, with respect to SOC and preferred terms by treatment group ( $Tables\ 3.2.1 - 3.2.3$ ).

If applicable, deaths (PT) will be included as part of AE/SAE analysis, including appropriate information such as date where available.

#### 7.5.6 Urine Drug Screening and Alcohol Breath Testing

Urine Drug Screening / Alcohol Breath Testing conducted during the study will be provided in a listing (*Listing 10.3*).



Protocol Nos.: PT010010 Date: 24 Aug 2017 

#### 7.5.7 Pregnancy Test

Pregnancy testing results conducted during the study will be provided in a listing (*Listing 10.4*).

#### 7.5.8 Prior/Concomitant Medications/Treatments

Prior and concomitant medications will be provided in listings (*Listing 10.1*). Information from both complete and partial dates will be utilized. Medications with end date of 'Ongoing' are considered concomitant. Should there not be sufficient information to determine whether a medication is prior or concomitant the status will be considered to be both prior and concomitant.

Concomitant medications and treatments will be summarized for the Safety Population, as well as presented by treatment group (*Table 1.5.1*). Frequency tables will present the frequency and proportion of subjects having received at least one concomitant medication during the course of the trial. Results will also be summarized with respect to subjects' receiving medications by coded preferred term.

#### 8. ANALYSES PERFORMED BEFORE DATABASE CLOSURE

Not applicable.

#### 9. CHANGES FROM METHODS PLANNED IN THE PROTOCOL

This SAP outlines the statistical methods for the display, summary and analysis of data collected within the scope of Pearl Therapeutics Inc. Protocol PT010010, Version 2.1 dated 15 Nov 2016.

# environment will be used for all statistical analyses. will be used for all PK parameter calculations. 11. REFERENCES



#### **APPENDIX 1: DATA HANDLING RULES**

STATISTICAL SOFTWARE

This appendix is provided in a separate document.

Protocol Nos.: PT010010 Date: 24 Aug 2017


## APPENDIX 2: TABLE OF CONTENTS FOR END-OF-TEXT TABLES, LISTINGS, AND FIGURES

#### 1 TABLES AND FIGURES

1.1 Summary of Subject Disposition, Demographics, and Baseline Characteristics

Table 1.1 Subject Disposition

(Analysis Set: All Subjects Screened)

Figure 1.1 Flow Chart of Subject Distribution

(Analysis Set: All Subjects Screened)

Table 1.2 Reasons for Withdrawal by Treatment

(Analysis Set: Safety Population)

Table 1.3 Analysis Populations by Treatment

(Analysis Set: All Subjects Randomized)

Table 1.4.1 Summary of Demographic Data by Treatment

(Analysis Set: Safety Population)

Table 1.4.2 Summary of Demographic Data by Treatment

(Analysis Set: PK Population)

Table 1.5.1 Summary of Concomitant Medications

(Analysis Set: Safety Population)

Table 1.6 Study Treatment Exposure and Compliance

(Analysis Set: Safety Population)

#### 1.2 Pharmacokinetic Data

Table 2.1.1 Descriptive Statistics for Plasma Concentrations of Budesonide (unit) by Treatment, Visit, and Timepoint

(Analysis Set: PK Population)
Protocol Nos.: PT010010 Date: 24 Aug 2017 

Figure 2.1.1 Mean (+/- SE) Plasma Budesonide Concentration-Time Profile after Single Dose Administration on Day 1 and Chronic Dose Administration on Day 8 (Linear-Linear Scale)

Analysis Set: PK Population

Figure 2.1.2 Mean Plasma Budesonide Concentration-Time Profile after Single Dose Administration on Day 1 and Chronic Dose Administration on Day 8 (Log-Linear Scale)

Analysis Set: PK Population

Table 2.1.2 Descriptive Statistics for Pharmacokinetic Parameters of Budesonide by Treatment and Visit

Analysis Set: PK Population

Table 2.2.1 Descriptive Statistics for Plasma Concentrations of Glycopyrronium (unit) by Treatment, Visit, and Timepoint

(Analysis Set: PK Population)

Figure 2.2.1 Mean (+/- SE) Plasma Glycopyrronium Concentration-Time Profile after Single Dose Administration on Day 1 and Chronic Dose Administration on Day 8 (Linear-Linear Scale)

Analysis Set: PK Population

Figure 2.2.2 Mean Plasma Glycopyrronium Concentration-Time Profile after Single Dose Administration on Day 1 and Chronic Dose Administration on Day 8 (Log-Linear Scale)

Analysis Set: PK Population

Table 2.2.2 Descriptive Statistics for Pharmacokinetic Parameters of Glycopyrronium by Treatment and Visit

Analysis Set: PK Population

Table 2.3.1 Descriptive Statistics for Plasma Concentrations of Formoterol (unit) by Treatment, Visit, and Timepoint

(Analysis Set: PK Population)

Figure 2.3.1 Mean (+/- SE) Plasma Formoterol Concentration-Time Profile after Single Dose Administration on Day 1 and Chronic Dose Administration on Day 8 (Linear-Linear Scale)

Analysis Set: PK Population





Protocol Nos.: PT010010 Date: 24 Aug 2017 

Figure 2.3.2 Mean Plasma Formoterol Concentration-Time Profile after Single Dose Administration on Day 1 and Chronic Dose Administration on Day 8 (/Log-Linear Scale)

Analysis Set: PK Population

Table 2.3.2 Descriptive Statistics for Pharmacokinetic Parameters of Formoterol by Treatment and Visit

Analysis Set: PK Population

Figure 2.4.1 Individual Plasma Concentration-Time Profile of Budesonide after Single Dose Administration on Day 1 and Chronic Dose Administration on Day 8 (Linear-Linear Scale)

(Analysis Set: PK Population)

Figure 2.4.2 Individual Plasma Concentration-Time Profile of Budesonide after Single Dose Administration on Day 1 and Chronic Dose Administration on Day 8 (Log-Linear Scale)

(Analysis Set: PK Population)

Figure 2.5.1 Individual Plasma Concentration-Time Profile of Glycopyrronium after Single Dose Administration on Day 1 and Chronic Dose Administration on Day 8 (Linear-Linear Scale)

(Analysis Set: PK Population)

Figure 2.5.2 Individual Plasma Concentration-Time Profile of Glycopyrronium after Single Dose Administration on Day 1 and Chronic Dose Administration on Day 8 (Log-Linear Scale)

(Analysis Set: PK Population)

Figure 2.6.1 Individual Plasma Concentration-Time Profile of Formoterol after Single Dose Administration on Day 1 and Chronic Dose Administration on Day 8 (Linear-Linear Scale)

(Analysis Set: PK Population)

Figure 2.6.2 Individual Plasma Concentration-Time Profile of Formoterol after Single Dose Administration on Day 1 and Chronic Dose Administration on Day 8 (Log-Linear Scale)

(Analysis Set: PK Population)

### 1.3 Safety Data

### 1.3.1 Adverse Events

Table 3.1.1 Summary of Subjects With At Least One Adverse Event


(Analysis Set: Safety Population)

Table 3.1.2 Summary of Treatment Emergent Adverse Events by System Organ Class and Preferred Term

(Analysis Set: Safety Population)

Table 3.2.1 Summary of Treatment Emergent Adverse Events by SOC, Preferred Term and Highest Severity – BGF MDI 320/14.4/9.6 µg

(Analysis Set: Safety Population)

Table 3.2.2 Summary of Treatment Emergent Adverse Events by SOC, Preferred Term and Highest Severity – BGF MDI  $160/14.4/9.6~\mu g$ 

(Analysis Set: Safety Population)

Table 3.2.3 Summary of Treatment Emergent Adverse Events by SOC, Preferred Term and Highest Severity –GFF MDI 14.4/9.6  $\mu g$ 

(Analysis Set: Safety Population)

### 1.3.2 Laboratory Data

Table 3.3.1 Summary of Laboratory Results by Time of Assessment – Hematology

(Analysis Set: Safety Population)

Table 3.3.2 Summary of Laboratory Results by Time of Assessment – Chemistry

(Analysis Set: Safety Population)

Table 3.3.3 Summary of Laboratory Results by Time of Assessment – Glucose and Potassium

(Analysis Set: Safety Population)

Table 3.3.4 Summary of Potentially Clinically Significant Laboratory Results Post-baseline – Glucose and Potassium

(Analysis Set: Safety Population)

Table 3.3.5 Summary of Laboratory Results by Time of Assessment – Urinalysis

(Analysis Set: Safety Population)

Table 3.3.6 All Potassium Records for Subjects with Newly Occurring or Worsening Potentially Clinically Significant Potassium Values Post-Baseline


Table 3.3.7 All Glucose Records for Subjects With Newly Occurring or Worsening Potentially Clinically Significant Glucose Values Post-Baseline

Table 3.3.8 All Records for Subjects With Newly Occurring or Worsening Potentially Clinically Significant Laboratory Values Post-Baseline Other Than Those for Glucose and Potassium

Table 3.3.9 Shifts from Baseline[a] to Day 8 Pre-Dose Laboratory Data – Hematology and Chemistry

(Analysis Set: Safety Population)

Table 3.3.9 Shifts from Baseline[a] to Day 8 Pre-Dose Laboratory Data – Hematology and Chemistry

(Analysis Set: Safety Population)

### 1.3.3 Vital Signs

Table 3.4.1 Summary of Vital Sign Measurements by Time of Assessment

(Analysis Set: Safety Population)

Table 3.4.2 Post-Baseline Potentially Clinically Significant Vital Sign Values

(Analysis Set: Safety Population)

Table 3.4.3 Listing of Potentially Clinically Significant Systolic and Diastolic Blood Pressure Increases and Decreases

(Analysis Set: Safety Population)

Table 3.4.4 Listing of Potentially Clinically Significant Tachycardia and Bradycardia Events

(Analysis Set: All Subjects Randomized)

### 2 DATA LISTINGS

### 2.1.1 Subject Disposition and Demographics

Listing 1.1 Listing of Subject Disposition and Demographic Data

(Analysis Set: All Subjects Screened)

Listing 1.2 Listing of Early Withdrawals by Trial Treatment

(Analysis Set: All Subjects Randomized)

### 2.1.2 Protocol Deviations


### Listing 2.1 Listing of Major Protocol Deviations

(Analysis Set: All Subjects Randomized)

Listing 2.2 Violation of Inclusion/Exclusion Criteria and Waivers

(Analysis Set: All Subjects Randomized)

### 2.1.3 Subjects Excluded from the Analysis Populations

Listing 3.1 Listing of Subjects Excluded From Analysis Populations

(Analysis Set: All Subjects Randomized)

### 2.1.4 Baseline Characteristics

Listing 4.1 Listing of Serology

(Analysis Set: All Subjects Randomized)

Listing 4.2 Listing of Medical and Surgical History

(Analysis Set: All Subjects Randomized)

### 2.1.5 Dosing and Compliance

Listing 5.1 Listing of Study Drug Dosing

(Analysis Set: All Subjects Randomized)

Listing 5.2 Compliance and Exposure to Study Treatment

(Analysis Set: All Subjects Randomized)

### 2.1.6 Adverse Events

Listing 7.1 Listing of Reported Adverse Events by Subject, SOC, Preferred Term and Onset Day

(Analysis Set: All Subjects Randomized)

Listing 7.2 Listing of Reported Serious Adverse Events by Subject, SOC, Preferred Term and Onset Day

(Analysis Set: All Screened Subjects)

### 2.1.7 Pharmacokinetic Data


Listing 8.1 Plasma Concentrations of Budesonide, Formoterol and Glycopyrronium by Treatment, Visit, Subject ID, and Timepoint

Analysis Set: PK Population

Listing 8.2 Derived Pharmacokinetic Parameters of Budesonide, Formoterol, and Glycopyrronium by Treatment/Visit and Subject ID

Analysis Set: PK Population

### 2.1.8 Laboratory Data

Listing 9.1 Listing of Laboratory Test Results - Hematology

(Analysis Set: All Subjects Randomized)

Listing 9.2 Listing of Laboratory Test Results - Chemistry

(Analysis Set: All Subjects Randomized)

Listing 9.3 Listing of Laboratory Test Results - Urinalysis

(Analysis Set: All Subjects Randomized)

### 2.1.9 Other Clinical Observations and Measurements

Listing 10.1 Listing of Reported Prior, Concomitant, and Post-Treatment Medication

(Analysis Set: All Subjects Randomized)

Listing 10.2 Listing of Vital Signs, Weight, and Height

(Analysis Set: All Subjects Randomized)

Listing 10.3 Listing of Urine Drug Screening / Alcohol Breath Testing

(Analysis Set: All Subjects Randomized)

Listing 10.4 Listing of Pregnancy Testing

(Analysis Set: All Subjects Randomized)

Listing 10.5 Listing of Comments

(Analysis Set: All Subjects Randomized)





Protocol Nos.: PT010010 Date: 24 Aug 2017 

## APPENDIX 3: CTCAE LABORATORY TEST CRITERIA FOR SHIFT TABLES AND CENTRAL LABORATORY REFERENCE RANGES FOR USE IN FLAGGING ABNORMAL VALUES

This appendix is provided in a separate document.




### **APPENDIX 1: DATA HANDLING RULES**

Programming of the tables, listings and figures will be performed using or a more recent version. The following table presents the algorithms to be used in to calculate the derived variables, including rules for handling other missing data or partial dates, or irregular/unexpected data issues.

| Category | | Description | Data Handling Rule |
|---|---|---|---|
| 1. | Age (years) | Age (years) | Age = integer part of ( [Informed Consent date – Birth date + 1]/365.25) |
| 2. | Smoking<br>History | Former smoker | Former smokers are defined as those who have stopped smoking for at least 6 months prior to Screening (Visit 1). |
| | | Months Since a Former<br>Smoker Quit | (Date of Screening Visit 1 – Date Former Smoker Quit)/30.4375. |
| 3. | Medical<br>History | Medical History Begin<br>Date of Condition | Begin date of condition will be imputed for all subjects as the 1 <sup>st</sup> of the month for the purpose of computing the onset day. |
| | Surgical<br>History | Surgical History Date of Surgery | Date of surgery will be imputed for all subjects as the 1 <sup>st</sup> of the month for the purpose of computing the onset day. |
| 5. | First and Last<br>Treatment<br>Dates | date/time of first and<br>last dose of a study<br>treatment | The date and time (24 hr. clock) of the first dose of study treatment will be taken from the Dosing eCRF. The date of the last dose of study treatment will be the last date of dosing from the Dosing eCRF for the treatment. |
| 6. | Last Visit<br>Date | Date of Last Visit | Date of last visit according to the Visit eCRF. |
| 7. | Last Study Participation Date (STDM variable, typically named RFPENDTC) | Last Study Participation Date (STDM variable, RFPENDTC), where SDTM denotes Study Data Tabulation Model | Last study participation date is defined as last known date of contact which would be the later of the following dates: last visit date, date of the last dose, date of last contact if lost-to-follow-up, date of telephone follow-up, or death date. |
| 8. | Study Day<br>Definitions | Study Day for<br>assessment/event which<br>occurs on or after the<br>start of study treatment | Study Day = Date of assessment/event – date of the first dose of study treatment + 1. |
| | | Study Day for assessments/events on | Study Day for assessments/events on days prior to the first dose of study treatment in the |



| <br> |
|---------------|

| Category | Description | Data Handling Rule |
|---|---|---|
| | days prior to the first<br>dose of study treatment<br>in the study | study |
| | Study Day Post-<br>Treatment of<br>Assessment or event<br>which occurs after<br>study treatment | Study Day = 'P' concatenated with the number of days post-treatment that the assessment or event occurred which is defined as Date of assessment/event – date of last dose of study treatment. |
| | Study Day of Randomization | Study Day of Randomization = date of randomization – date of the first dose of study treatment in the study + 1. Study Day is 1 if baseline day is on the day of randomization. |
| | First Dose Day | <b>First Dose Day</b> in the study is defined as the study day of the first dose of study treatment in the study (Study Day 1). |
| | Last Dose Day | Last Dose Day in the study is defined as the study day of the last dose of study treatment in the study (defined as the last date of dosing from the Dosing CRF pages). |
| | Last Study Day | For subjects who did not receive study treatment in the study (e.g., Non-Randomized subjects), Last Study Day is defined as (the later of the last visit date and the date of last contact for subjects lost-to-follow-up from the Study Completion/Early Discontinuation CRF) — Date of Screening Visit + 1. For subjects who received study treatment in the study, Last Study Day is defined as (the later of the last visit date and the date of last contact for subjects lost-to-follow-up from the Study Completion/Early Discontinuation CRF) — first dose date in the study + 1. |
| | Days Since Last Dose for event (e.g., Death) | Days Since Last Dose is defined as date of event – date of last dose of study treatment. |
| O Duration of | The duration of any event | The duration of any event is defined as (stop date – start date + 1). |
| 9. Duration of event | The duration of any event | The duration of any event is defined as (stop date – start date + 1). |




| Category | Description | Data Handling Rule |
|---|---|---|
| 10. Multiple assessments for the same visit | Vital Signand Laboratory assessments | <ul> <li>All data will be listed in data listings.</li> <li>The last of multiple valid assessments within a post-baseline study time window will be used for summaries and statistical testing.</li> <li>If there are multiple laboratory values for the same parameter at post-baseline predose of a visit, the last value will be chosen for analysis.</li> <li>The mean of all available pre-dose vital sign measurements for a vital sign parameter taken prior to the start of dosing for the Treatment Period will be used for calculation of baseline for a parameter.</li> </ul> |
| 11. Special Lab Value Handling (not including PK values) | Lab values with a prefix such as: '>', '<', '+' and 'Less than' Etc. | <ul> <li>'&gt;': use the available original value +0.001 in the analyses.</li> <li>'&lt;': use the available original value -0.001 in the analyses.</li> <li>'+': use the available original value without the prefix in the analyses.</li> <li>'&gt;=': use the available original value in the analyses.</li> <li>'&lt;=': use the available original value in the analyses.</li> </ul> |
| 12. Prior. concomitant, and post- treatment medication / treatment | Prior, concomitant, and post-treatment medication/treatment | 1. Prior medication/treatment: is any medication/treatment taken prior to the first dose of study medication in the study (or the date of the randomization visit, Visit 3, if the date of the start of study medication is missing), even if this medication/treatment continued into the study medication treatment period. A medication/treatment will be considered prior if the start date of the medication/treatment is missing or the medication/treatment start date is before |



| _ |
|-------|

| Category | Description | Data Handling Rule |
|---|---|---|
| | | first dose date of study medication in the study (or the date of the randomization visit, Visit 3, if the date of the start of study medication is missing). 2. A medication/treatment will be identified as a concomitant medication/treatment if any of the following are true: O The start date is on or after the date of the start of study treatment (or the date of randomization, Visit 3, if missing), but prior to the date of completion of study medication (for subjects not having discontinued treatment early) or the date of discontinuation of study medication (for subjects who discontinued treatment early). O The end date is prior to the date of completion of study medication (for subjects not having discontinued treatment early) or the date of the discontinuation of study medication (for subjects who discontinued treatment early), but the end date is on or after the start of study medication in the study (or the date of the randomization visit, Visit 3, if missing). The medication/treatment is checked as 'Ongoing', and the start date of the medication/treatment is prior to the date of completion of study medication (for subjects not having discontinued treatment early) or the date of the discontinuation of study medication (for subjects not having discontinued treatment early) or the date of the discontinuation of study medication (for subjects not having discontinued treatment early) or the date of the discontinuation of study medication (for subjects who discontinued treatment early). |
| | | the date of completion of study medication (for subjects not having discontinued |



Date: 24 August 2017


| Category | Description | Data Handling Rule |
|---|---|---|
| | | treatment early) or on or after the date of discontinuation of study medication (for subjects who discontinued treatment early) will not be considered concomitant, but will be considered a <b>Post-Treatment medication</b> . 4. Any medication/treatment which cannot be identified as Prior, Concomitant, or Post-Treatment will be considered as being in each of the possible categories depending on available information |
| 13. Adverse event | Missing severity | For the AE summary by severity, an AE with missing severity will be deemed as Severe. Imputed values will not be listed in data listings. |
| | Missing relationship to study drug | For AE summary by relationship, an AE with a missing relationship to study drug will be deemed as Definitely related. Imputed values will not be listed in data listings. |
| | Treatment-emergent adverse event | An adverse event is considered treatment- emergent if an event occurs (or if there was a worsening [intensity and/or severity changed to worsened grades]) after the first dose of randomized study medication and on or before the date of discontinuation from or completion of randomized study medication. An adverse event that begins on the same date as the first dose of randomized study medication is treatment-emergent if the AE begins after the time of first dose or if the time of AE onset is unknown. A non-serious adverse event will not be considered to be treatment-emergent if its date of onset is after the date of completion of study medication (for subjects not having discontinued treatment early) or after the date of discontinuation from study medication (for subjects who discontinued treatment early). An SAE will not be considered to be treatment- emergent if its date of onset is after the date of completion of study medication (for subjects |



|-------|---|----|----|

| Category | Description | Data Handling Rule |
|---|---|---|
| | | <ul> <li>not having discontinued treatment early) or after the date of discontinuation from study medication (for subjects who discontinued treatment early).</li> <li>If the AE start date is partial/missing, then</li> <li>If AE start date is completely missing, then the AE is considered as treatment-emergent.</li> <li>If both AE start month and day are missing and AE start year is the same or after the first dose year, then the AE is considered as treatment-emergent.</li> <li>If AE start day is missing and AE start year and month are the same or after the first dose year and month, then the AE is considered as treatment-emergent.</li> <li>Missing/incomplete (partial) AE start and end</li> </ul> |
| 14. Treatment Duration | Treatment Duration | dates will not be imputed for data listings. Treatment duration is defined as Date of last dose of a study treatment - Date of first dose of a study treatment +1. |
| 15. Total Years of Exposure | Total years of exposure to study treatment | Total exposure (years) for a treatment as a whole is defined as the sum of all days of exposure for a treatment /365.25. |
| 16. Exposure (days) | Exposure (days) | Exposure is defined as (Date of the last dose of the study treatment – Date of first dose of the study treatment + 1). |
| 17. Total Expected Puffs | Total expected number of puffs taken of a study treatment | The expected number of puffs for a test day which is the first date of treatment or the last date of treatment will be 2, the expected number of puffs for the last date of treatment which is not a test day will be 4 when a PM dose has been taken and then 2 otherwise, and the expected number of puffs on dates after the first date of treatment and prior to the last date of treatment will be 4. Thus, for test treatments, the total expected number of puffs will be 4 x (treatment end date – treatment start |



|-------|---|----|----|

| Category | Description | Data Handling Rule |
|---|---|---|
| | | date-1) + expected number of puffs on last day of treatment + expected number of puffs on first day of treatment. |
| 18. Treatment Compliance (%) | Treatment Compliance (%) for a treatment | Percent compliance is defined as (total number of puffs of study treatment taken on a study day/total expected puffs taken on a study day) averaged across all days of a subject's dosing between start of study treatment and last day on study treatment) x 100. For MDI test treatments, the expected number of puffs for a test day which was the first or the last date of treatment is 2, the expected number of puffs for the last date of treatment which was not a test day is 4 when a PM dose was taken and then 2 otherwise; the expected number of doses on dates after the first date of treatment and prior to the last date of treatment is 4. |
| 19. Hard coding | Hard coding for data analysis | Hard Coding is not allowed during data analysis unless if agreed in writing by the Sponsor. |
| 20. PK analysis | Considerations to be made in the calculation of AUC and $\lambda_z$ and for descriptive statistics | <ul> <li>The following considerations will be made in the calculation of AUC and λ<sub>z</sub> and descriptive statistics:</li> <li>AUC will be calculated by the linear-log trapezoidal method</li> <li>The final selection of samples for calculation of λ<sub>z</sub> will be based on visual inspection of individual log-concentration-time profiles.</li> <li>The time range of samples used to estimate λ<sub>z</sub> should preferably exceed the derived terminal half-life t<sub>½</sub> (= ln 2/λ<sub>z</sub>). This consideration may affect the interpretability of the estimated λ<sub>z</sub> and t<sub>½</sub>.</li> <li>All the samples used to calculate λ<sub>z</sub> should ideally fall in the log-linear elimination phase. PK modeling may</li> </ul> |



Date: 24 August 2017


| Category | Description | Data Handling Rule |
|---|---|---|
| | | <ul> <li>be used as a complementary tool to determine the start of the elimination phase, i.e., where the decline in plasma concentration is mainly due to elimination.</li> <li>At least three samples above LLQ obtained during the log-linear elimination phase will be included in the calculation of the λ<sub>z</sub>. If there are not at least three samples above the LLQ in the log linear elimination phase, λ<sub>z</sub> will not be estimated.</li> <li>All values below LLQ will be ignored (set to missing) in the noncompartmental analysis for computing pharmacokinetic parameters except that Day 1 pre-dose concentrations below the LLQ will be set to 0. For descriptive statistics for concentrations and for the concentration figures, all values below LLQ will be assigned a value of ½ LLQ except for Day 1 predose which will be assigned a value of 0 (no geometric mean will be calculated for Day 1 pre-dose).</li> </ul> |

BGF MDI PT010010

Version 1.0 24 August 2017 

CTCAE LABORATORY TEST CRITERIA FOR SHIFT TABLES AND CENTRAL LABORATORY REFERENCES RANGES FOR USE IN FLAGGING ABNORMAL VALUES APPENDIX 3

Trial Sponsor: Pearl Therapeutics, Inc.

**Protocol Number:** PT010010-01

Budesonide, Glycopyrronium, and Formoterol Fumarate Inhalation Aerosol Investigational Drug:

(PT010, BGF metered dose inhaler [MDI])

Glycopyrronium and Formoterol Fumarate Inhalation Aerosol

(PT003, GFF MDI)

Indication: COPD

Drug Number: PT010

**Dosage Form/Strength:** • BGF MDI 320/14.4/9.6 µg ex-actuator BID

BGF MDI 160/14.4/9.6 μg ex-actuator BID

GFF MDI 14.4/9.6 μg ex-actuator BID

**Protocol Title:** A Phase I, Randomized, Double-Blind, Parallel-Group, Study to Assess the Pharmacokinetics and Safety of Two Doses of PT010 and a Single Dose of PT003 in Healthy Chinese Adult Subjects Following A Single Administration and After Chronic

Administration for 7 Days


# CTCAE LABORATORY TEST CRITERIA

| Investigations | | | | |
|---|---|---|---|---|
| | | Grade | ıde | |
| Adverse Event | 1 | 2 | 3 | 4 |
| Alanine | >ULN - 3.0 x ULN | >3.0 – 5.0 x ULN | >5.0 – 20.0 x ULN | >20.0 x ULN |
| aminotransferase | | | | |
| increased | | | | |
| Alkaline phosphatase | >ULN $- 2.5 x$ ULN | >2.5-5.0 x ULN | >5.0-20.0 x ULN | >20.0 x ULN |
| increased | | | | |
| Aspartate | >ULN - 3.0 x ULN | >3.0 - 5.0 x ULN | >5.0 – 20.0 x ULN | >20.0 x ULN |
| aminotransferase | | | | |
| increased | | | | |
| Blood bilirubin | >ULN - 1.5 x ULN | >1.5-3.0 x ULN | >3.0 – 10.0 x ULN | >10.0 x ULN |
| increased | | | | |
| Cholesterol high | >ULN $-300 mg/dL;$ | >300 – 400 mg/dL; >7.75 | >400-500 mg/dL; | >500 mg/dL;>12.92 |
| | >ULN -7.75 mmol/L | -10.34 mmol/L | >10.34 –12.92 mmol/L | mmol/L |
| Creatinine increased | >1-1.5 x baseline; | >1.5-3.0 x baseline; | >3.0 baseline; $>3.0 - 6.0$ | NTN x 0.9< |
| | >ULN -1.5 x ULN | >1.5 - 3.0 x ULN | xULN | |
| Chloride | | | | |
| GGT increased | >ULN - 2.5 x ULN | >2.5 – 5.0 x ULN | >5.0 – 20.0 x ULN | >20.0 x ULN |
| Hematocrit | n/a | n/a | n/a | n/a |


| Investigations | | | | |
|---|---|---|---|---|
| | | Grade | de | |
| Adverse Event | 1 | 2 | 3 | 4 |
| Hemoglobin increased | Increase in $>0-2$<br>gm/dL above ULN or<br>above baseline if<br>baseline is above | Increase in >2 – 4 gm/dL<br>above ULN or above<br>baseline if baseline is<br>above ULN | Increase in >4 gm/dL<br>above ULN or above<br>baseline if baseline is<br>above ULN | n/a |
| Anemia (hemoglobin<br>decreased) | Hemoglobin (Hgb) <lln-10g <lln-100="" <lln-6.2="" dl;="" g="" l;="" l<="" mmol="" td=""><td>Hgb &lt;10.0 – 8.0 g/dL;<br/>&lt;6.2 – 4.9 mmol/L;<br/>&lt;100 – 80g/L</td><td>Hgb &lt;8.0 g/dL; &lt;4.9 mmol/L; &lt;80 g/L; transfusion indicated</td><td>Life-threatening consequences; urgent intervention indicated</td></lln-10g> | Hgb <10.0 – 8.0 g/dL;<br><6.2 – 4.9 mmol/L;<br><100 – 80g/L | Hgb <8.0 g/dL; <4.9 mmol/L; <80 g/L; transfusion indicated | Life-threatening consequences; urgent intervention indicated |
| Serum Iron | n/a | n/a | n/a | n/a |
| Ferritin | n/a | n/a | n/a | n/a |
| Red blood cells<br>(erythrocytes) | n/a | n/a | n/a | n/a |
| Leukocytosis (White blood cell increased) (a) | n/a | n/a | >100,000/mm³ | Clinical manifestations of leucostasis; urgent intervention indicated |


| Investigations | | | | |
|---|---|---|---|---|
| | | Grade | ıde | |
| Adverse Event | 1 | 2 | 3 | 4 |
| White blood cell decreased | <pre><lln -="" 3000="" mm³;<="" pre=""><lln -="" 10°="" 3.0="" l<="" pre="" x=""></lln></lln></pre> | $<3000-2000/\text{mm}^3;$<br>$<3.0-2.0 \times 10^9/\text{L}$ | <2000 – 1000/mm <sup>3</sup> ; $<$ 2.0 – 1.0 x 10 <sup>9</sup> /L | $<1000/\text{mm}^3;$<br>$<1.0 \times 10^9 / \text{L}$ |
| White blood cell differential | n/a | n/a | n/a | n/a |
| Platelet count<br>decreased | <pre><lln -="" 10<sup="" 75,000="" 75.0="" <lln="" mm3;="" x="">9/L</lln></pre> | <75,000 50,000/mm3;<br><75.0 - 50.0 x 10°/L | <50,000 – 25,000/mm3;<br><50.0 – 25.0 x 10 <sup>9</sup> /L | <25,000/mm3;<br><25.0 x 10°/L |
| Mean corpuscular<br>volume | n/a | n/a | n/a | n/a |
| Mean cell hemoglobin<br>(MCH) | n/a | n/a | n/a | n/a |
| MCH concentration | n/a | n/a | n/a | n/a |

BGF MDI PT010010

| Metabolism and Nutrition Di | Disorders | | | |
|---|---|---|---|---|
| | | 9 | Grade | |
| Adverse Event | 1 | 2 | 3 | 4 |
| Acidosis | pH <normal, but="">=7.3</normal,> | 1 | pH <7.3 | Life-threatening consequences |
| Alkalosis | pH>normal, but <=7.5 | 1 | pH>7.5 | Life-threatening consequences |
| Urea | n/a | n/a | n/a | n/a |
| Blood Urea Nitrogen (BUN) | n/a | n/a | n/a | n/a |
| Proteinuria | 1+ proteinuria;<br>urinary protein<br><1.0g/24 hrs | Adults: 2+ proteinuria; urinary protein 1.0 – 3.4 g/24 hrs. Pediatric: urin P/C (protein/creatinine) ratio 0.5 - 1.9 | Adults: urinary protein >=3.5 g/24 hrs; Pediatric: urine P/C >1.9 | n/a |
| Hypercalcemia | Corrected serum calcium of >ULN - 11.5 mg/dL; >ULN - 2.9 mmol/L; Ionized calcium >ULN - 1.5 mmol/L | Corrected serum calcium of >11.5 - 12.5 mg/dL; >2.9 - 3.1 mmol/L; Ionized calcium >1.5 - 1.6 mmol/L; symptomatic | Corrected serum calcium of >12.5 - 13.5 mg/dL; >3.1 - 3.4 mmol/L; lonized calcium >1.6 - 1.8 mmol/L; hospitalization indicated | Corrected serum calcium of >13.5 mg/dL; >3.4 mmol/L; Ionized calcium >1.8 mmol/L; life-threatening consequences |


| Metabolism and Nutrition Di | sorders | | | |
|---|---|---|---|---|
| | | 9 | Grade | |
| Adverse Event | 1 | 2 | 3 | 4 |
| Hyperglycemia | Fasting glucose value > ULN - 160 | Fasting glucose value >160 - 250 | >250 - 500 mg/dL; >13.9<br>- 27.8 mmol/L; | >500 mg/dL; >27.8 mmol/L; life- |
| | mg/dL; Fasting glucose value >ULN | mg/dL; Fasting<br>glucose value >8.9 - | hospitalization indicated | threatening<br>consequences |
| Hyperkalemia | >ULN - 5.5 mmol/L | >5.5 - 6.0 mmol/L | >6.0 - 7.0 mmol/L; | >7.0 mmol/L; life- |
| (Potassium Increased) | | | hospitalization indicated | threatening consequences |
| Hypermagnesemia (Magnesium Increased) | >ULN - 3.0 mg/dL; | n/a | >3.0 - 8.0 mg/dL; >1.23 - | >8.0 mg/dL; >3.30 |
| | mmol/L | | | threatening |
| | | | | consequences |
| Hypernatremia (Sodium | >ULN - 150 mmol/L | >150 - 155 mmol/L | >155 - 160 mmol/L; | >160 mmol/L; life- |
| moreased) | | | nospitalization mulcated | consequences |
| Hypertriglyceridemia | 150 mg/dL - 300<br>mg/dL; 1.71 mmol/L | >300 mg/dL - 500<br>mg/dL; >3.42 | >500 mg/dL - 1000<br>mg/dL; >5.7 mmol/L - | >1000 mg/dL;<br>>11.4 mmol/L; life- |
| | - 3.42 mmol/L | mmol/L - 5.7 | 11.4 mmol/L | threatening |
| | | mmol/L | | consequences |
| Hypoalbuminemia (Albumin | <lln -="" 3="" dl;<="" g="" td=""><td>&lt;3 - 2 g/dL; &lt;30 -</td><td>&lt;2 g/dL; &lt;20 g/L</td><td>Life-threatening</td></lln> | <3 - 2 g/dL; <30 - | <2 g/dL; <20 g/L | Life-threatening |
| Decreased) | ~LLIN = 30 g/L | 70 g/L | | urgent intervention |
| | | | | indicated |


| Metabolisin and Mutition Disorders | | | | |
|---|---|---|---|---|
| | | ) | Grade | |
| Adverse Event | 1 | 2 | 3 | 4 |
| Hypocalcemia (Calcium | Corrected serum | Corrected serum | Corrected serum calcium | Corrected serum |
| Loci casou) | 8.0 mg/dL; <lln -<="" td=""><td>7.0 mg/dL; &lt;2.0 -</td><td><pre><!-- < '.0 - 0.0 mg/dz,</pre--></pre></td><td>mg/dL: &lt;1.5</td></lln> | 7.0 mg/dL; <2.0 - | <pre><!-- < '.0 - 0.0 mg/dz,</pre--></pre> | mg/dL: <1.5 |
| | 2.0 mmol/L; Ionized | 1.75 mmol/L; | Ionized calcium <0.9-0.8 | mmol/L;Ionized |
| | calcium <lln -="" 1.0<="" td=""><td>Ionized calcium</td><td>mmol/L;</td><td>calcium &lt;0.8</td></lln> | Ionized calcium | mmol/L; | calcium <0.8 |
| | mmol/L | <1.0- 0.9 mmol/L; | hospitalizationindicated | mmol/L;life- |
| | | symptomatic | | threatening |
| | | | | conseduences |
| Hypoglycemia (Glucose | <lln -="" 55="" dl;<="" mg="" td=""><td>&lt;55 - 40 mg/dL;</td><td>&lt;40 - 30 mg/dL; &lt;2.2 -</td><td>&lt;30 mg/dL; &lt;1.7</td></lln> | <55 - 40 mg/dL; | <40 - 30 mg/dL; <2.2 - | <30 mg/dL; <1.7 |
| Decreased) | <pre><lln -="" 3.0="" l<="" mmol="" pre=""></lln></pre> | <3.0 - 2.2 mmol/L | 1.7 mmol/L | mmol/L; life- |
| | | | | threatening |
| | | | | consequences; |
| | | | | seizures |
| Hypokalemia (Potassium | <pre><lln -="" 3.0="" l<="" mmol="" pre=""></lln></pre> | <lln -="" 3.0<="" td=""><td>&lt;3.0 - 2.5 mmol/L;</td><td>&lt;2.5 mmol/L; life-</td></lln> | <3.0 - 2.5 mmol/L; | <2.5 mmol/L; life- |
| Decreased) | | mmol/L; | hospitalization indicated | threatening |
| | | symptomatic; | | consequences |
| | | intervention<br>indicated | | |
| Hypomagnesemia | <lln -="" 1.2="" dl;<="" mg="" td=""><td>&lt;1.2 - 0.9 mg/dL;</td><td>&lt;0.9 - 0.7 mg/dL; &lt;0.4 -</td><td>&lt;0.7 mg/dL; &lt;0.3</td></lln> | <1.2 - 0.9 mg/dL; | <0.9 - 0.7 mg/dL; <0.4 - | <0.7 mg/dL; <0.3 |
| (Magnesium Decreased) | <lln -="" 0.5="" l<="" mmol="" td=""><td>&lt;0.5 - 0.4 mmol/L</td><td>0.3 mmol/L</td><td>mmol/L; life-</td></lln> | <0.5 - 0.4 mmol/L | 0.3 mmol/L | mmol/L; life- |
| | | | | threatening |
| | | | | consequences |
| Hyponatremia (Sodium | <lln -="" 130="" l<="" mmol="" p=""></lln> | n/a | <130 - 120 mmol/L | <120 mmol/L; life- |
| Decreased) | | | | threatening |
| | | | | consequences |


| Metabolism and Nutrition Di | Disorders | | | |
|---|---|---|---|---|
| | | ) | Grade | |
| Adverse Event | 1 | 2 | 3 | 4 |
| Hypophosphatemia<br>(Phosphate Decreased) | <pre><lln -="" 2.5="" dl;<="" mg="" td=""><td>&lt;2.5 - 2.0 mg/dL;<br/>&lt;0.8 - 0.6<br/>mmol/L</td><td><pre>&lt;2.0 - 1.0 mg/dL; &lt;0.6 - mmol/L; = 0.3 mmol/L life- threatening consequences</pre></td><td><pre>&lt;1.0 mg/dL; &lt;0.3 mmol/L; life- threatening consequences</pre></td></lln></pre> | <2.5 - 2.0 mg/dL;<br><0.8 - 0.6<br>mmol/L | <pre>&lt;2.0 - 1.0 mg/dL; &lt;0.6 - mmol/L; = 0.3 mmol/L life- threatening consequences</pre> | <pre>&lt;1.0 mg/dL; &lt;0.3 mmol/L; life- threatening consequences</pre> |

| Renal and Urinary Disorders | | | | |
|---|---|---|---|---|
| | | 9 | Grade | |
| Adverse Event | 1 | 2 | 3 | 4 |
| Chronic kidney disease | eGFR (estimated Glomerular Filtration Rate) or CrCl (creatinine clearance) <lln -60="" 1.73="" m<sup="" min="" ml="">2 or proteinuria 2+ present; urine protein/creatinine &gt;0.5</lln> | eGFR or CrCl 59 -<br>30 ml/min/1.73 m <sup>2</sup> | eGFR or CrCl 29 - 15<br>ml/min/1.73 m <sup>2</sup> | eGFR or CrCl <15<br>ml/min/1.73 m²;<br>dialysis or renal<br>transplant indicated |


| Acute kidney injury | Creatinine level increase of >0.3 mg/dL; creatinine 1.5 - 2.0 x above baseline | Creatinine 2 – 3 x above baseline | Creatinine >3 x baseline or >4.0 mg/dL; hospitalization indicated | Life-threatening consequences; organ failure; urgent operative intervention indicated |
|---|---|---|---|---|
| (a) Grade 1 and Grade 2 r<br>(LabCorp) | not categorized in CTCAE | 4; Grade 1 and 2 based o | a) Grade 1 and Grade 2 not categorized in CTCAE4; Grade 1 and 2 based on reference laboratory alert criteria of 40,000 /mm³ LabCorp) | riteria of 40,000 /mm³ |

Version 1.0 24 August 2017


## Protocol Reference Range Definitions

For reference range definitions, refer to the document pt010010 lab range site 001 20170405.pdf